CLINICAL TRIAL: NCT02620332
Title: Multiple Islet Peptide Administration in Type 1 Diabetes (MultiPepT1De)
Acronym: MultiPepT1De
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MultiPep001
Record Dates: First submitted 2015-09-24; First posted 2015-12-03 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo injection (Placebo Comparator): Water for injection
  Interventions: Other: Placebo
- MultiPepT1De injection low dose (Experimental): Mix of peptides administered once a month over a period of 20 weeks (6 injections in total)
  Interventions: Drug: MultiPepT1De injection
- MultiPepT1De injection medium dose (Experimental): Mix of peptides administered once a month over a period of 20 weeks (6 injections in total)
  Interventions: Drug: MultiPepT1De injection
- MultiPepT1De injection high dose (Experimental): Mix of peptides administered once a month over a period of 20 weeks (6 injections in total)
  Interventions: Drug: MultiPepT1De injection

INTERVENTIONS:
Drug: MultiPepT1De injection — A mix of peptides
  Other Names: Multipeptide injection
  Arms: MultiPepT1De injection high dose; MultiPepT1De injection low dose; MultiPepT1De injection medium dose
Other: Placebo — Water for injection
  Arms: Placebo injection

SUMMARY:
Type 1 diabetes is an autoimmune disease in which the insulin secreting βcells of the pancreas are destroyed such that the patient is reliant on injection of insulin to adequately control blood glucose levels for the remainder of his/her life. The autoimmune process targets proteins in beta-cells which are termed autoantigens. This is a Phase 1 study using a novel investigational medicinal product (IMP) known as MultiPepT1De in a study of safety and tolerability of administration in patients with recent onset Type 1 diabetes. MultiPepT1De is a mixture of peptides from islet auto antigens. The mixture has been designed to induce or restore immunological tolerance to the beta-cell and thus control or limit autoimmunity to protect beta-cells

DETAILED DESCRIPTION:
Recent onset type 1 diabetes patients will be randomized into 4 groups of 6 subjects and each group will receive 6 injections of either placebo, low, medium or high dose of IMP; each injection is intradermal and spaced 1 month apart.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Type 1 diabetes
* Age 18-45 years
* Maximum of 4 years from diagnosis
* Evidence of ≥1 autoantibody against β-cell autoantigens
* Possession of the HLA-DR4 (DRB1*0401) genotype
* Residual β-cell function (peak C-peptide >200)

Exclusion Criteria:

* Females who are pregnant, breast-feeding or not using adequate forms of contraception.
* Use of β-cell stimulants, immunosuppressive or immunomodulatory therapies, including systemic steroids within 1 month prior to randomization, any monoclonal antibody therapy given for any indication and any antigen-specific

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-10-20 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2018-04-06 (Actual)

PRIMARY OUTCOMES:
Assessment of MultiPepT1De safety profile | Every 28 days for 147 days
  Safety assessed through measurement and comparison of any reactions or hypersensitivity to MultipepT1De injection vs placebo. Number of adverse events will also be compared between groups with the addition of safety monitoring blood tests

SECONDARY OUTCOMES:
Assessment of residual beta cell function and markers of metabolic control | 24 weeks versus baseline
  Measured by a change in stimulated C-peptide production, daily insulin usage, glycated haemoglobin levels and amplitude of glucose excursions from baseline and between groups
Assessment of T lymphocyte immune response to islet cell antigens | 24 weeks versus 12 weeks
  Comparison of changes in antigen specific T lymphocyte responses longitudinally following peptide treatment and versus placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jake Powrie, MD FRCP, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust; Mark Peakman, MBBS PhD, Study Director — King's College London
Locations (1):
- Guy's Hospital, London, United Kingdom

REFERENCES:
- [Derived] Liu YF, Powrie J, Arif S, Yang JHM, Williams E, Khatri L, Joshi M, Lhuillier L, Fountoulakis N, Smith E, Beam C, Lorenc A, Peakman M, Tree T. Immune and Metabolic Effects of Antigen-Specific Immunotherapy Using Multiple beta-Cell Peptides in Type 1 Diabetes. Diabetes. 2022 Apr 1;71(4):722-732. doi: 10.2337/db21-0728. PMID 35073398